CLINICAL TRIAL: NCT04334499
Title: Investigation of the Relationship Between Mitochondrial DNA in Vitreous Fluid and Blood in Patients With Eye Disease or Ocular Trauma.
Brief Title: Mitochondrial DNA in Vitreous Fluid and Blood in Patients With Eye Disease or Ocular Trauma.
Status: Withdrawn | Type: Observational
Why Stopped: The study was never initiated; Principal Investigator determined that it was not feasible to continue with the study at this time.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0291
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Eye Diseases; Ophthalmic Trauma; Mitochondrial DNA; Age Related Macular Degeneration; Glaucoma; Diabetic Retinopathy
Keywords: mitochondrial DNA; opthalmic trauma; age related macular degeneration; glaucoma; inflammation; inflammatory marker; diabetic retinopathy
MeSH Terms: conditions — Eye Diseases; Macular Degeneration; Glaucoma; Diabetic Retinopathy; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of vitreous humor and plasma will be collected for analysis of mtDNA by RTq-PCR.
  Remaining samples will be maintained in a de-identified state for unidentified future research without additional consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Age Related Macular Degeneration: Subjects with Age Related Macular Degeneration upon evaluation for ocular surgery that may involve the discard of vitreous humor tissue.
  Interventions: Other: Sample collection from tissue discard
- Glaucoma: Subjects with Glaucoma upon evaluation for ocular surgery that may involve the discard of vitreous humor tissue.
  Interventions: Other: Sample collection from tissue discard
- Diabetic Retinopathy: Subjects with Diabetic Retinopathy upon evaluation for ocular surgery that may involve the discard of vitreous humor tissue.
  Interventions: Other: Sample collection from tissue discard
- Ocular Trauma: Subjects with Ocular Trauma upon evaluation for ocular surgery that may involve the discard of vitreous humor tissue.
  Interventions: Other: Sample collection from tissue discard
- Control: Subjects with no ocular disease or trauma comorbidities upon evaluation for ocular surgery that may involve the discard of vitreous humor tissue.
  Interventions: Other: Sample collection from tissue discard

INTERVENTIONS:
Other: Sample collection from tissue discard — Collection of vitreous humor tissue and venous blood from subjects undergoing ocular surgery that may provide vitreous humor discarded tissue.

SUMMARY:
This study is to characterize mitochondrial DNA (mtDNA) populations in adults with eye injuries and eye diseases. The eye exam is often hindered by the clouding of tissues involved in injury or disease. This protocol examines the use of mtDNA populations as indicators of developing inflammation and resolution of injury. This may be used to provide proactive treatment or define appropriate treatment needs beyond the indications of an ophthalmological exam.

DETAILED DESCRIPTION:
The study aim to test correlation between the presence of the mitochondrial DNA in vitreous fluid and blood in patients that are admitted to UTMB's Eye clinic. The goal of the study is to analyze 4 groups of 30 samples of each major ocular disease and injury: age-related macular degeneration, glaucoma and diabetic retinopathy and ocular trauma. Up to 300 subjects may be consented to this study in order to meet recruitment goals. In this study we will use only otherwise discarded eye's vitreous together with a blood sample that is collected during surgery. Patients with ophthalmic surgery scheduled that may result in discarded vitreal fluid will be identified from the clinic schedule or by physician in the emergency room. The possibility of vitreous collection in a surgery may be uncertain. If a subject does not have discarded vitreous from a given surgery they will be screen failed prior to blood draw or data collection from electronic medical record from that moment forward. Subjects will be approached when appropriate for interest in participation in the study by their clinical faculty surgeon. An informed consent briefing will be provided by the clinical research coordinator with an opportunity to ask questions of both the coordinator, the clinical faculty surgeon and the principle investigator. Copies of the consent will be provided for the patient to take home. Additional opportunity for questions the morning of surgery will be provided. Consent signature will be obtained prior to any medication administration the upon admission for surgery. Samples if available will be collected during the eye surgery. Up to 1ml of vitreous fluid and up to 10 ml of blood will be collected from each patient. Samples will be stored at room temperature and transferred directly to Dr. Szczesny's laboratory. Vitreous fluid will be frozen for further analysis and blood plasma will be processed using histopaque and centrifugation prior freezing. Two types of analysis will be conducted with collected biospecimens.1) Total DNA will be isolated, follow by analysis with real-time quantitative polymerase chain reaction (RTq-PCR) using set of primers to identify the presence of the mitochondrial DNA and nuclear DNA as a control. 2) Extracellular vesicles will be isolated using ultracentrifugation or commercially available kit followed by analysis of the mitochondrial and nuclear DNA and/or plasma membrane markers using RTq-PCR and/or Western blot. Electronic medical records will be accessed to collect demographics and ophthalmologic diagnostic information and information on other comorbidity diagnoses.

These data points will include age in years, gender, race, ethnicity, presence of age related macular degeneration(AMD) (y/n), type and stage of AMD, use of AREDs vitamins, treatments of AMD, Glaucoma(y/n), type and stage of glaucoma, diabetes, blood glucose, diabetic retinopathy (y/n), type and stage of diabetic retinopathy, treatments of diabetic retinopathy and amount of time prior to this planned surgery, hypertension type and stage, renal disease type and stage, smoking history, cancer, cancer type, treatment or surgery, viral diagnoses (HIV, CMV, HCV), blunt eye trauma history, cataract history, lens removal surgery, cause of vitrectomy, concomitant medications and procedures, eye exam observations relevant to inflammatory processes, Optical coherence tomography data. IOP, visual field [VF] data, visual acuity, gonioscopic findings,.

ELIGIBILITY:
Inclusion Criteria:

* a) Target group

  1. Age ≥ 20 years old
  2. Subjects must not be nursing, pregnant or planning to become pregnant. Subjects of child bearing potential must have a documented negative pregnancy test at the time of preoperative assessment or not be of child bearing potential. Identified eye disease including but not limited to age-related macular degeneration, glaucoma and/or diabetic retinopathy.
  3. Scheduled ophthalmic surgery with expected vitreal humor discard.
  4. Subject has provided written informed consent to participate in this protocol. b) Control group

  <!-- -->

  1. Age ≥ 20 years old
  2. Subjects must not be nursing, pregnant or planning to become pregnant. Subjects of child bearing potential must have a documented negative pregnancy test at the time of preoperative assessment or not be of child bearing potential.
  3. Lack of identified eye disease.
  4. Scheduled ophthalmic surgery with expected vitreal humor discard.
  5. Subject has provided written informed consent to participate in this protocol.

Exclusion Criteria:

* a) Target group

  1. Age < 20 years old
  2. Subject is nursing, pregnant, planning to become pregnant or of child bearing potential and does not agree to the use of reliable method of contraception during their participation in the study. A pregnancy test must be administered to women of childbearing potential at the time of preoperative assessment.
  3. Identified eye disease including but not limited to age-related macular degeneration, glaucoma and/or diabetic retinopathy.
  4. Subject has not completed informed consent to participate in this protocol. b) Scheduled ophthalmic surgery with expected vitreal humor discard Control group

  <!-- -->

  1. Age < 20 years old
  2. Subject is nursing, pregnant, planning to become pregnant or of child bearing potential and does not agree to the use of reliable method of contraception during their participation in the study. A pregnancy test must be administered to women of childbearing potential at the time of preoperative assessment.
  3. Lack of identified eye disease.
  4. Subject has not completed informed consent to participate in this protocol. Scheduled ophthalmic surgery with expected vitreal humor discard.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects suffering eye disease or ocular trauma and healthy subjects undergoing ocular surgery which may include the discard of vitreous humor.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Quantitation of mitochondrial DNA in vitreous humor and serum samples | 1 day
  mtDNA quantitation by RTq-PCR

SECONDARY OUTCOMES:
Evaluation of mtDNA quantitation versus ocular comorbidities as described in electronic medical record. | 1 month
  Collection of comorbidity data from electronic medical record and comparison with quantiative analysis of mtDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Szczesny, Ph.D., Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No
Study records will be kept confidential as required by law. Except when required by law, your identifiers will not be disclosed outside of the University of Texas Medical Branch (UTMB). For records disclosed outside of UTMB, you will be assigned a unique code number. The key to this code will be kept in a password protected encrypted format on a limited access server behind the UTMB firewall. It will be destroyed at the end of data collection for this study.
  Study samples will also be kept in a de-identified state with the same 4 digit code as the data collection. These samples will be maintained in secured laboratories of the Department of Ophthalmology. The de-identified samples may be maintained past the end of the study for future research without additional consent. Future researchers will have no information on the identity of the subjects.